CLINICAL TRIAL: NCT04706494
Title: A Randomized, Double-blind, Placebo-controlled, Cross-over Study to Investigate the Efficacy of an Acute Dose of AlphaWave® LTheanine on Stress in a Healthy Adult Population
Brief Title: A Study to Investigate the Efficacy of AlphaWave® L-Theanine on Stress
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ethical Naturals, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 19LSHE
Record Dates: First submitted 2020-02-12; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AlphaWave® LTheanine (Experimental)
  Interventions: Dietary Supplement: AlphaWave® LTheanine
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AlphaWave® LTheanine — 200 mg of AlphaWave® LTheanine
  Arms: AlphaWave® LTheanine
Dietary Supplement: Placebo — microcrystalline cellulose
  Arms: Placebo

SUMMARY:
AlphaWave® L-theanine will be compared against placebo to evaluate how the investigational study product effects on salivary cortisol, EEG readings, blood pressure, and heart rate in a moderately stressed and otherwise healthy adult population. It is hypothesized that participants taking the AlphaWave® L-theanine will have reduced stress levels as assessed by the parameters stated. Participants will be consuming the investigational study product or placebo in the clinic only.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age, inclusive
* BMI between 18.5 to 29.9 kg/m2, inclusive
* Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, total endometrial ablation) or have been post-menopausal for at least 1 year prior to screening OR,
* Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

  * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
  * Double-barrier method
  * Intrauterine devices
  * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
  * Vasectomy of partner at least 6 months prior to screening
* Individuals with moderate stress as determined by the Perceived Stress Scale (scores ranging from 14 - 26 are considered moderate stress)
* Have a regular sleep-wake cycle with a bedtime between 9:00 pm and 12:00 am and receive between 7 and 9 hours of sleep for at least 3 weeks prior to baseline
* Agrees to maintain current sleep schedule throughout study
* Agrees to maintain current levels of diet, supplements, and exercise until the end of the study
* Agrees to refrain from exercising 24-hours prior to the visits
* Agrees to abstain from using hair products on the day of visits
* Willingness to complete questionnaires, records, diaries associated with the study, and to complete all clinic visits
* Healthy as determined by medical history, laboratory results, and physical exam as assessed by the QI

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Clinically significant abnormal laboratory results at screening as assessed by the QI
* Participants who have a known allergy to the test material's active or inactive ingredients
* Current employment that calls for rotating shift work or shift work that will disrupt normal circadian rhythm or have worked shift work in the last 3 weeks
* Travelled across 1 or more time zones in the last 3 weeks and/or is anticipating more travel
* Self reported epilepsy and/or seizures
* Type I or Type II Diabetes
* Unstable metabolic disease or chronic diseases as assessed by the QI
* Current or history of any significant disease of the gastrointestinal tract
* Hypertension treated with medication or supplements or untreated hypertension
* Self reported anxiety or depression
* Significant cardiovascular event in the past 6 months as assessed by the QI
* Major surgery in the past 3 months or individuals who have planned surgery during the course of the trial. Participants with minor surgery will be considered on a case-by-case basis by the QI
* Individuals with an autoimmune disease or are immune-compromised
* History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones symptom-free for 6 months
* Self reported current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
* Self reported confirmation of medical or neuropsychological condition and/or cognitive impairment that, in the QI's opinion, could interfere with study participation
* Self reported blood/bleeding disorders that will have an effect on safety outcomes as assessed by the QI
* Alcohol or drug abuse within the last 12 months
* High alcohol intake (>2 standard drinks per day)
* Use of medicinal cannabinoid products
* Chronic use of cannabinoid products (>2 times/week). Occasional use to be assessed by the QI on a case by case basis
* Use of tobacco and nicotine-containing products within 60 days of baseline
* Current use of prescribed medications listed: antibiotics, antiepileptics, antiseizure medications, sedatives, hypnotics
* Current use of over-the-counter medications, supplements, foods, and/or drinks listed: caffeine, green tea, L-theanine supplements, melatonin supplements, valerian root supplements, GABA supplements, tart cherries/drinks/supplements, amla, ashwagandha, rhodiola, shatavari, ginseng
* Blood donation 30 days prior to screening or a planned donation 30-days of the last study visit
* Participants in a clinical research trial within 30 days of screening
* Individuals who are unable to give informed consent
* Any other condition that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
The change in salivary cortisol levels from pre- to post-tests between AlphaWave® LTheanine versus placebo. | 9 days
  Assessed by analysis of saliva sample at baseline and end of study
The change in EEG total alpha wave readings from pre- to post-tests between AlphaWave® LTheanine versus placebo. | 9 days
  Measured and analyzed at baseline and end of study
The change in EEG frontal alpha wave readings from pre- to post-tests between AlphaWave® LTheanine versus placebo. | 9 days
  Measured and analyzed at baseline and end of study
The change in EEG midline theta wave readings from pre- to post-tests between AlphaWave® LTheanine versus placebo. | 9 days
  Measured and analyzed at baseline and end of study

SECONDARY OUTCOMES:
The change in heart rate from pre-to post-test between the investigational product versus placebo | 9 days
  Measured at baseline and end of study
The change in blood pressure from pre- to post-test between the investigational product versus placebo | 9 days
  Measured at baseline and end of study
The change in State-Trait Anxiety Inventory (STAI) from pre- to post-test between the investigational product versus placebo | 9 days
  Assessed by the participants' answers to the questionnaire
The change in Visual Analog Scale (VAS) from pre- to post-tests between the investigational product versus placebo | 9 days
  Assessed by the participants' answers to the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mal Evans, PhD, Study Chair — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evans M, McDonald AC, Xiong L, Crowley DC, Guthrie N. A Randomized, Triple-Blind, Placebo-Controlled, Crossover Study to Investigate the Efficacy of a Single Dose of AlphaWave(R) L-Theanine on Stress in a Healthy Adult Population. Neurol Ther. 2021 Dec;10(2):1061-1078. doi: 10.1007/s40120-021-00284-x. Epub 2021 Sep 25. PMID 34562208